CLINICAL TRIAL: NCT00384644
Title: Skeletal Muscle Oxygenation in Critically Ill
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Matej Podbregar, UMC Ljubljana
Other Study IDs: NIRS-1
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Heart Failure; Sepsis; Septic Shock; Cardiogenic Shock
Keywords: heart failure; sepsis; septic shock; cardiogenic shock
MeSH Terms: conditions — Heart Failure; Sepsis; Shock, Septic; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: sepsis, septic shock ptients
  Interventions: Device: NiRS measurment of tissue oxygenation
- 2: cardiogenic shock patients
  Interventions: Device: NiRS measurment of tissue oxygenation

INTERVENTIONS:
Device: NiRS measurment of tissue oxygenation — NiRS measurment of tissue oxygenation

SUMMARY:
It is possible to measure skeletal muscle tissue oxygenation (StO2) using near infrared spectroscopy(NIRS). It is performed non invasively. We want to compare usually used invasive methods for assessing adequacy of flow to StO2 in critically ill. Aim is to faster and non invasively estimate adequacy of flow to make therapeutic algorithms efficient.

DETAILED DESCRIPTION:
Introduction

The duration and severity of tissue hypoxia have been related to increased mortality. Maintenance of adequate oxygen delivery (DO2) is essential to preserve organ function, as a sustained low DO2 is a path to organ failure and death. DO2 does not have influence on oxygen consumption (VO2) until it reaches critically low values (DO2crit), when VO2 starts to fall. Low cardiac output states (cardiogenic, hypovolemic and obstructive types of shock), anemic and hypoxic hypoxemia are characterized by a decreased DO2 but preserved oxygen extraction ratio (OER=the ratio of DO2 to VO2, VO2/ DO2) so that DO2crit remains normal. In distributive shock, the oxygen extraction capability is altered so that the critical oxygen extraction ratio is typically decreased. These situations are typically associated with an increased DO2crit, and VO2 can become dependant on DO2 even when the latter is normal or elevated. These observations help to characterize the four principal types of circulatory shock, however this classification is somewhat simplistic as several types of alternations may coexist, in particular in cardiogenic shock. Rhodes et al. reported that outcome was more favorable in septic patients whose VO2 increased after dobutamine administration. DO2 also increased in survivors. On the other hand DO2 did not increase in patients whose VO2 did not increase. In dobutamine test proposed by Rhodes et al. the hemodynamic response was influenced by cardiovascular reserve and the degree of stimulation of adrenoreceptors at baseline. Unfortunately global measurements of DO2 and VO2 may not be sensitive enough to be clinically relevant. They may fail to detect regional perfusion abnormalities as in splanchnic circulation.

Measurement of mixed venous oxygen saturation (SvO2) from the pulmonary artery is used for the calculations of the VO2 and has been advocated as an indirect index of tissue of tissue oxygenation and prognostic predictor in critically ill patients. Catheterization of pulmonary artery is costly, has inherent risks and its usefulness remains under debate. Not surprisingly the monitoring of central venous oxygen saturation (ScvO2) was suggested as a simpler and chipper assessment of global DO2 to VO2 ratio.

Near infrared spectroscopy (NIRS) is a technique for continuous, non-invasive, bedside monitoring of tissue oxygen saturation (StO2). Like pulse oximetry, NIRS uses the principles of light transmission and absorption to non-invasively measure the concentrations of oxygenated hemoglobin and reduced hemoglobin in tissue. NIRS offers greater tissue penetration and does not discriminate between compartments. Therefore it provides a global assessment of oxygenation in all vascular compartments (arterial, venous and capillary) in sample volume of underlining tissue. We have previously shown that thenar muscle tissue oxygen saturation during stagnant ischemia decreases slower in septic shock patients compared to patients with severe sepsis, localized infection and healthy volunteers. This may be due to microcirculatory or metabolic changes, and probably correlates to muscle tissue oxygen consumption. The rate of StO2 decrease correlated with SOFA score, norepinephrine requirement, and plasma lactate concentration. As recently described, StO2 in sample volume of underlining tissue depends in vivo on 3 major determinants: the concentration in oxy-hemoglobin, capillary recruitment and the vascular size (vasodilatation or constriction). The StO2 during stagnant ischemia has then to be viewed in light of these determinants. The gradual decrease (slope) of StO2 after cuff inflation-induced vascular occlusion depends mainly on the augmentation of the concentration of deoxy-hemoglobin and estimates tissue oxygen consumption and to a lesser degree on vessel de-recruitment. The StO2 upslope during reperfusion (cuff deflation) can be analyzed in light of flow papers during ischemia/reperfusion test. Vasodilatation after ischemia leads to recruitment of more vessels and increase in the local blood flow, which in turn results in a StO2 increase. It remains unclear which of the described changes is more influential, however this StO2 increase mirrors the maximal local DO2 at the time of measurement. The development on NIRS signal processing might be able to provide a clinical important tissue hemoglobin concentration index and local oxygen consumption as shown by De Blasi et al., such an index may help to clarify the mechanism(s) by which StO2 signal varies.

The aim of our study was to study skeletal muscle oxygen kinetics in low flow state due to combined cardiogenic and septic circulatory failure, relate it with central heamodynamic variables and outcome. We hypothesized that basal StO2 could relate to ScvO2, because blood flowing through upper limb muscles importantly contributes to flow through superior vena cava. The second hypothesis was that decrease of skeletal muscle OER and lower muscle oxygen consumption are more pronounced in patients with septic component of circulatory failure due to microcirculatory and metabolic changes seen in sepsis, what results in higher mortality.

MATERIALS AND METHODS

Patients Study protocol was approved by the National Ethics Committee of Slovenia, informed consent was obtained from all patients or their relatives. Study was performed during October 2004 and January 2006. After initial hemodynamic resuscitation, transthoracic ultrasound heart examination was performed in all patients admitted to our ICU. In patients with primary heart disease, low cardiac output, and no signs of hypovolemia, a right heart catheterization with a pulmonary artery floating catheter (PAFC)(Swan-Ganz CCOmboV CCO/SvO2/CEDV, Edwars Life Sciences, USA) was performed after decision of treating physician. The site of insertion was confirmed by the transducer waveform, the length of catheter insertion and chest radiography. In all patients systemic arterial pressure was measured invasively using radial or femoral arterial catheterization. Patients with inserted PAFC and signs of low flow state (cardiac index less then 3.0 L/min/m2) were included in our study. PAFC data were calculating using standard formula.

Localized infection, severe sepsis and septic shock were defined according to ACCP/SCCM consensus conference definitions (1992). All patients received standard treatment of localized infection, severe sepsis and septic shock including: source control, fluid infusion, catecholamine infusion, organ failure replacement and/or support therapy, intensive control of blood glucose and corticosteroid substitution therapy. Mechanically ventilated patients were sedated with midazolam and/or propofol infusion and no paralytic agents were used.

Measurements

Skeletal Muscle Oxygen Kinetics

Thenar muscle StO2 was measured non-invasively by NIRS (15mm Probe, InSpectra™, Hutchinson Technology Inc., USA). The values were continuously monitored and stored into a computer using InSpectra ™ software. The StO2 was monitored before, during and after upper arm ischemia-reperfusion test (UIRT) which was standardized as follows: a rapid cuff inflation above elbow towards 260 mmHg to stop flow and to induce a decrease in StO2 for 90 seconds, cuff deflation with continuous measurement of StO2 increase, overshooting and stabilization. Measurements were performed immediately after PAFC insertion (in first 24 to 72 hours after admission), the second measurement was performed 12-24 hours after the first measurement, the third measurement was performed (only if patient was still alive and still had PAFC inserted) in 48 hours after the first measurement. In spontaneously breathing patients and healthy volunteers measurements were performed after 15 minutes of bed rest, avoiding any muscular contractions.

In figure 1 schematic StO2 measurement line-drawing during UIRT is presented. The following parameters were obtained: basal StO2 (%): basal StO2 before cuff inflation (maximal thenar muscle StO2 was found by moving probe over thenar prominence); StO2 downslope during cuffing (∆downStO2)%/sec); StO2 upslope (∆upStO2)%/sec) after cuffing release; overshootStO2 (%): maximal StO2 after cuffing release. Inspectra measures content of hemoglobin in sample volume of underlining tissue - Tissue Haemoglobin Index (THI). Average of muscle THI before and at the end of cuff inflation was reported. These data were automatically obtained using the Inspectra Analysis Program V2.0 (Hutchinson Technology Inc., USA) running in MatLab 7.0 (MathWorks Inc., USA). Estimation of muscle oxygen consumption (mVO2Nirs) and muscle oxygen extraction ratio (mOER) were calculated using the following formulas:

mVO2Nirs= ΔdownStO2 * THI* (-1), mOER(%)= (1- basalStO2/overshootStO2)* 100.

Severity of disease Sepsis-related Organ Failure Assessment (SOFA score) was calculated at the time of each measurement to asses the level of organ dysfunction. Dobutamine, norepinephrine requirement represented the dose of drug during the Sto2 measurement. Used of levosimendan is reported if patient received the drug less then a week before inclusion in the study. Use of intra-aortic balloon pump during ICU stay is reported.

Laboratory analysis Blood was withdrawn from superior vena cava approximately 2cm above right atrium and pulmonary artery was performed at the time of each StO2 measurement to determine ScvO2 (%) and SvO2(%) respectively. In view of the known problems arising during sampling from pulmonary artery, including the possibility of contaminating artery blood with pulmonary capillary blood, all samples from this site were withdrawn over 30s, using a low-negative pressure technique, and never with the balloon inflated . A standard volume of 1mL of blood was obtained from each side after withdrawn of dead-space blood and flushing fluid. All measurements were made using a cooximeter (RapidLab 1265, Bayer HealthCare, Germany).

Plasma lactate concentration was measured using enzymatic colorimetric method (Lactate, Roche Diagnostics, Germany) at the time of each StO2 measurement.

Data analysis StO2 curves were analyzed by Inspectra Analysis Program V2.0. Linear regression was used to extrapolate the rate of Δdown- and Δup- StO2 during UIRT. Data was expressed as median ± standard deviation (SD). Non parametric test: Kolmogorov-Smirnov, Wilcoxon and Fisher exact test were used (SPSS 10.0 for Windows ™, SPSS Inc., USA). Spearman correlation test was used to determine correlation. To compare muscle tissue StO2 variables during UIRT, ScvO2 and SvO2: bias, systemic disagreement between the measurements (mean difference between two measurements), and precision, the random error in measuring (standard deviation of bias), were calculated. The limits of agreement were arbitrary set by Bland and Altman as the bias± 2 SD. To determine the variables independently associated with survival uni- and multivariate logistic regression (Forward Stepwise (Likelihood Ratio)) was used. The p value of <0.05 (2-tailed) was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* all typs of shock (cardiogenic, septic, hypovolemic, obstractive)

Exclusion Criteria:

* patients/relatives refuse to participate in study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Intensive care patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2004-04; Primary Completion 2009-01 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matej Podbregar, MD PhD, Principal Investigator — Medical Faculty, University of Ljubljana
Locations (1):
- Clinical Center Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Background] Pareznik R, Knezevic R, Voga G, Podbregar M. Changes in muscle tissue oxygenation during stagnant ischemia in septic patients. Intensive Care Med. 2006 Jan;32(1):87-92. doi: 10.1007/s00134-005-2841-8. Epub 2005 Nov 1. PMID 16261341
- [Derived] Mozina H, Podbregar M. Near-infrared spectroscopy during stagnant ischemia estimates central venous oxygen saturation and mixed venous oxygen saturation discrepancy in patients with severe left heart failure and additional sepsis/septic shock. Crit Care. 2010;14(2):R42. doi: 10.1186/cc8929. Epub 2010 Mar 23. PMID 20331856
- [Derived] Podbregar M, Mozina H. Skeletal muscle oxygen saturation does not estimate mixed venous oxygen saturation in patients with severe left heart failure and additional severe sepsis or septic shock. Crit Care. 2007;11(1):R6. doi: 10.1186/cc5153. PMID 17227587